CLINICAL TRIAL: NCT00003624
Title: A Limited Access Trial Using Amifostine for Protection Against Cisplatin and 3-Hour Paclitaxel-Induced Neurotoxicity
Brief Title: Amifostine in Treating Women With Ovarian, Peritoneal, Cervical, Fallopian Tube, Uterine, or Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Supportive Care
Other Study IDs: CDR0000066705; GOG-9805
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2006-05

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Neurotoxicity; Ovarian Cancer; Primary Peritoneal Cavity Cancer; Sarcoma
Keywords: stage I cervical cancer; stage II cervical cancer; stage III cervical cancer; stage IV cervical cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial adenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; neurotoxicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Neurotoxicity Syndromes; Ovarian Neoplasms; Sarcoma; Carcinoma, Ovarian Epithelial | interventions — Amifostine; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of amifostine in reducing the risk of side effects caused by cisplatin and paclitaxel in treating women who have ovarian, peritoneal, cervical, fallopian tube, uterine, or endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of amifostine in reducing significant peripheral neuropathy in women with ovarian, peritoneal, cervical, fallopian tube, uterine, or endometrial cancer treated with cisplatin and paclitaxel. II. Determine the proportion of patients on this regimen who experience significant peripheral neuropathy 3 months after completing chemotherapy. III. Assess the overall toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 3 hours, amifostine IV over 10 minutes, and cisplatin IV over 90 minutes. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Neurotoxicity is assessed and vibration perception threshold testing is performed prior to each course of chemotherapy and at 3 months following the last treatment. Patients are followed every 3 months for 2 years, then every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 29-59 patients will be accrued for this study within 18-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Ovarian, primary peritoneal, cervical, or fallopian tube carcinoma, uterine sarcoma, or endometrial adenocarcinoma for which the proposed treatment is cisplatin plus paclitaxel Must be ineligible for a higher priority GOG protocol

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-3 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No hypertension for which medication cannot be discontinued for 24 hours through the day of each chemotherapy treatment Other: No history of neuropathy (e.g., diabetic neuropathy) No significant infection Prior malignancy allowed if disease free for at least 12 months No physical disabilities precluding vibration perception threshold testing of the upper and lower extremity (e.g., amputation, paraplegia)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for ovarian, primary peritoneal, or fallopian tube carcinoma, uterine sarcoma, or endometrial adenocarcinoma Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy except for cervical carcinoma Surgery: Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-12; Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Moore, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (8):
- United States (8):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Cleveland Clinic Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Moore DH, Donnelly J, McGuire WP, Almadrones L, Cella DF, Herzog TJ, Waggoner SE; Gynecologic Oncology Group. Limited access trial using amifostine for protection against cisplatin- and three-hour paclitaxel-induced neurotoxicity: a phase II study of the Gynecologic Oncology Group. J Clin Oncol. 2003 Nov 15;21(22):4207-13. doi: 10.1200/JCO.2003.02.086. PMID 14615449